CLINICAL TRIAL: NCT06652490
Title: Short-axis/out-of-plane Approach Versus Oblique- Axis Approach for Ultrasound-guided Internal Jugular Venous Catheterization in Infants.
Brief Title: Short-axis/out-of-plane Approach Versus Oblique- Axis Approach for US Guided IJV Catheterization in Infants.
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS60/2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-22 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-02

CONDITIONS: Central Line Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A (control group): ( n=25 ): CVL insertion in the right internal jugular vein using ultrasound. The US probe is placed perpendicular to the venous anatomy in the SAX approach.
  Interventions: Procedure: Short-axis/out-of-plane approach versus oblique- axis approach for ultrasound-guided internal jugular venous catheter.
- Group B (comparative group): ( n=25 ): CVL insertion in the right internal jugular vein using ultrasound. The US probe is aligned at 45° angulation clockwise with the venous anatomy in the OAX approach.
  Interventions: Procedure: Short-axis/out-of-plane approach versus oblique- axis approach for ultrasound-guided internal jugular venous catheter.

INTERVENTIONS:
Procedure: Short-axis/out-of-plane approach versus oblique- axis approach for ultrasound-guided internal jugular venous catheter. — In the group A, The US probe will be placed perpendicular to the venous anatomy in the SAX approach.
  In the group B, The US probe will be aligned at 45° angulation with the venous anatomy, and combined with an in plane needle insertion technique. The needle will be advanced from lateral to medial.

SUMMARY:
The investigators will measure and compare the rate of acute complications, success rate, number of attempts to successful cannulation between ultrasound-guided short axis approach and oblique axis approach during internal jugular venous catheterization in infants.

DETAILED DESCRIPTION:
1. pre-procedure settings: The history will be obtained from patient's parents. Investigations will be checked to all patients as (complete blood picture and coagulation profile) to avoid coagulopathy and thrombocytopenia.

   All patients will be attached to standard monitoring (blood pressure (non-invasive), heart rate, and pulse oximetry).

   Groups:

   Patients will be assigned randomly by using a computer -generated table of random numbers into two groups:
   * Group A (control group): ( n=25 ): CVL insertion in the right internal jugular vein using ultrasound. The US probe is placed perpendicular to the venous anatomy in the SAX approach.
   * Group B (comparative group): ( n=25 ): CVL insertion in the right internal jugular vein using ultrasound. The US probe is aligned at 45° angulation?clockwise with the venous anatomy in the OAX approach.
2. procedure Settings: Monitor will be connected and pulse oximetry (SPO2), baseline non-invasive blood pressure (NIBP), heartrate (HR), electrocardiogram (ECG) will be obtained.

In this study, we will use US machine with small linear probe with frequency 5 - 10 Hz and the procedure will be held by the most senior Anaesthesiologist experience in pediatric central venous catheterization for at least 3 years.

The procedure will be held under aseptic condition, Using US, after GA in OR, the anatomical location and patency of the IJV will be assessed with the patient placed in the Trendelenburg position, with the head slightly rotated to the contralateral side. With all sterile precautions, a 4 french introducer needle mounted on a syringe is inserted into the IJV guided by real time US imaging. Once blood is freely aspirated, the US probe is set aside and the syringe removed from the needle. Then the guide wire will be advanced through the needle into the vessel and the catheter will be advanced using the Seldinger technique after guidewire position is confirmed with US. The guidewire will be then removed. Using US, placement of the catheter in the vein will confirmed following which the catheter will be secured in place using sutures. The position of the CVC wiil be also confirmed by a chest radiograph at the end of the procedure.

In the group A, The US probe will be placed perpendicular to the venous anatomy in the SAX approach.

In the group B, The US probe will be aligned at 45° angulation with the venous anatomy, and combined with an in plane needle insertion technique. The needle will be advanced from lateral to medial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 12 months
* Physical status: patients requiring CVC in their management

Exclusion Criteria:

* patient's parents refuse to do the study
* Coagulopathy (INR > 1.5, platelets count < 50.000), use of anti-coagulant or anti platelet therapy) (Sunny et al, 2022)
* Infection, wounds or subcutaneous hematoma close to the puncture site
* history of previous surgical intervention at the cannulation site
* subcutaneous emphysema, penetrating neck trauma or cervical trauma

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will be carried out on infants who require central venous access through IJV as part of their management in operating room (OR) if they consented to be part of the study from their parents.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Difference in the rate of acute complications between the two groups. | Post-procedure, through study completion (average 1 year)
  acute complications as posterior venous wall puncture (PVWP) (ultrasonographic identification of the needle tip or guidewire at any site deeper than the posterior wall of the IJV during cannulation attempts), skin and subcutaneous hematoma, arterial puncture (any pulsatile blood reflux through the needle observed during the procedure), pneumothorax, hemothorax and catheter misplacement (catheter tip identified at any place other than the superior vena cava in the control chest radiograph)

SECONDARY OUTCOMES:
Difference in the rate of first successful cannulation attempt. | Post procedure, through study completion (average 1 year)
  first successful cannulation attempt (successful venous puncture and successful smooth insertion of guidewire from the first needle puncture without withdrawal of the needle)
the flash time. | Post procedure, through study completion (average 1 year)
  time to completion flash time (The time interval between skin puncture and observing blood at the syringe hub)
the number of needle redirection. | Post procedure, through study completion (average 1 year)
  number of needle redirection (redirection of the needle without complete withdrawal of the needle)
unsuccessful cannulation. | Post procedure, through study completion (average 1 year)
  unsuccessful cannulation (a cannulation is considered unsuccessful if it had to be performed using an approach that differed from that to which the patient had been initially chosen for and also if the operator was unable to cannulate the vein within 3 attempts)

CONTACTS AND LOCATIONS:
Overall Officials: Engy Y Attallah, M.B.B.C.H, Principal Investigator — Anesthesia resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All dana will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2025
Access Criteria: Free